CLINICAL TRIAL: NCT00342563
Title: Treatment With Mecamylamine in Smoking and Non-smoking Alcohol Dependent Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26364
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Alcoholism
Keywords: mecamylamine; treatment; alcohol dependence; smoking
MeSH Terms: conditions — Alcoholism; Smoking | interventions — Mecamylamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Mecamylamine- Smoker (Experimental)
  Interventions: Drug: mecamylamine
- Placebo-Smoker (Placebo Comparator)
  Interventions: Drug: Placebo
- Mecamylamine- Non-Smoker (Experimental)
  Interventions: Drug: mecamylamine
- Placebo-Non-Smoker (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mecamylamine — mecamylamine 10mg/day
  Arms: Mecamylamine- Non-Smoker; Mecamylamine- Smoker
Drug: Placebo — Placebo
  Arms: Placebo-Non-Smoker; Placebo-Smoker

SUMMARY:
The purpose of the study will be to evaluate the efficacy of mecamylamine in reducing alcohol consumption in smoking and non-smoking alcohol dependent patients.

We hypothesize that mecamylamine will result in a greater reduction of alcohol consumption than placebo. We further hypothesize that mecamylamine will be effective in reducing both alcohol consumption and smoking in a subset of alcoholics who also smoke.

DETAILED DESCRIPTION:
RESEARCH PLAN: Although there are two FDA approved medications for the treatment of alcohol dependence (naltrexone and disulfiram), the robust efficacy of both compounds in reducing alcohol consumption has recently been called into question. Given the high rates of alcohol dependence among the general population, development and testing of novel medications is of great importance.

Mecamylamine, a noncompetitive NACh receptor antagonist has been shown to be useful in smoking cessation when used in combination with transdermal nicotine. To our knowledge, clinical studies examining the effectiveness of mecamylamine in alcoholism have not been conducted. However, there is evidence from animal research that mecamylamine can block the effects of alcohol. Infusion of mecamylamine into the ventral tegmental area antagonized ethanol-induced dopamine release in rats. More importantly, mecamylamine decreased alcohol intake and preference in alcohol-preferring rats. In two studies with healthy volunteers mecamylamine was effective in attenuating the euphoric effects of alcohol and reducing the craving for alcohol.

This is the first study designed to test the clinical efficacy of mecamylamine in a sample of alcohol dependent patients who either do or do not smoke.

For the proposed project we will recruit 60 treatment seeking patients between the ages of 18 and 60 who meet criteria for alcohol dependence and may or may not smoke. Patients will be randomized into two groups (30 patients in each group): one dose of mecamylamine (10mg) or placebo in a double-blind fashion for 12 weeks. Patients will be asked to come for follow up 3 months after completing the study. Patients will be excluded if they: take medications thought to influence drinking behavior, have a significant underlying medical conditions, such as cerebral, renal, thyroid, hepatic or cardiac pathology; have a history of glaucoma, prostatic hypertrophy, urethral obstruction, cerebral arteriosclerosis, pyloric stenosis, or a history of hypersensitivity to mecamylamine; or meet current criteria for Bipolar Disorders, Schizophrenia and Schizophrenia-type Disorders, Major Depression or Posttraumatic Stress Disorders (PTSD). Females who are pregnant or lactating will also be excluded.

We hypothesize that mecamylamine will result in a greater reduction of alcohol consumption than placebo among the alcohol dependent patients. We further hypothesize that mecamylamine will be effective in reducing both alcohol consumption and smoking in a subgroup of alcoholics who also smoke.

ELIGIBILITY:
Inclusion Criteria:

* individuals with DSM-IV diagnosis of alcohol dependence
* smokers and non-smokers
* patients who do not require psychotropic medication for the management of their psychiatric symptoms
* individuals with a history of substance dependence (other than alcohol and tobacco) but have not met criteria for substance dependence in the past 30 days
* women with acceptable method of contraception

Exclusion Criteria:

* pregnant women
* medications thought to influence drinking behavior including: acamprosate, disulfiram, naltrexone and ondansetron
* underlying medical conditions
* history of glaucoma, prostatic hypertrophy, urethral obstruction, cerebral arteriosclerosis, pyloric stenosis, or a history of hypersensitivity to mecamylamine
* DSM-IV diagnosis of bipolar disorder, schizophrenia, and schizophrenia-type disorders
* unstable medical conditions
* patients who require psychotropic medication for the management of an active psychiatric disorder
* patients on pharmacological treatment for alcohol and/or nicotine dependence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2004-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismene Petrakis, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Gandelman E, Petrakis I, Kachadourian L, Ralevski E. Negative Affect Intensity and Hostility in Individuals With Alcohol Use Disorder With or Without Posttraumatic Stress Disorder. J Dual Diagn. 2018 Apr-Jun;14(2):96-101. doi: 10.1080/15504263.2018.1434264. Epub 2018 Apr 25. PMID 29461925

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mecamylamine- Smoker | Mecamylamine Non-Smoker | Placebo Smoker | Placebo Non-Smoker
Started | 41 | 27 | 40 | 28
Completed | 35 | 19 | 26 | 22
Not Completed | 6 | 8 | 14 | 6

BASELINE CHARACTERISTICS:
Population: One hundred and thirty six (136) individuals were randomized in this study with equal number of participants assigned to treatment (n=68) and placebo (n=68) groups. Randomization was stratified by gender and smoking status.
Groups:
- Mecamylamine-Smoker: mecamylamine: mecamylamine 10mg/day
- Total: Total of all reporting groups
Arm/Group | Mecamylamine-Smoker | Mecamylamine-Non-Smoker | Placebo-Smoker | Placebo- Non-Smoker | Total
Number analyzed (Participants) | 41 | 27 | 40 | 28 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.83 (8.42) | 50.93 (9.55) | 47.28 (8.69) | 51.14 (10.28) | 48.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 6 | 4 | 20
  Male | 35 | 23 | 34 | 24 | 116
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 17 | 14 | 18 | 18 | 67
  White | 23 | 13 | 21 | 10 | 67
  Other | 1 | 0 | 1 | 0 | 2
Veteran Status [Number; unit: participants]
  Veteran | 19 | 9 | 18 | 8 | 54
  Non-Veteran | 22 | 18 | 22 | 20 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percent Heavy Drinking Days During Active Treatment Phase
Description: Data were calculated as number of heavy drinking days (heavy drinking days is defined as 5 drinks on a single occasion for men and 4 for women) average during 90 days of treatment.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: days
Groups:
- Mecamylamine- Smokers; Mecamylamine- Non-Smoker: mecamylamine: mecamylamine 10mg/day
- Placebo-Smoker: Placebo
Arm/Group | Mecamylamine- Smokers | Mecamylamine- Non-Smoker | Placebo-Smoker | Placebo- Non-Smoker
Number analyzed (Participants) | 41 | 27 | 40 | 28
days | 16.75 (4.33) | 24.28 (5.30) | 20.51 (4.57) | 21.78 (5.11)

2. Primary Outcome: Self-report Weekly Craving Via Obsessive Compulsive Drinking Scale (OCDS)
Description: The OCDS is a 14-item (rated 0-4), self-administered questionnaire for characterizing and quantifying the obsessive and compulsive cognitive aspects of craving and heavy (alcoholic) drinking, such as drinking-related thought, urges to drink, and the ability to resist those thoughts and urges. A higher total score indicates higher craving and ranges from 0-48.
Time Frame: 12 weeks
Population: Scores presented are total, and then by subgroup.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mecamylamine | Placebo
Number analyzed (Participants) | 68 | 68
units on a scale
  Total | 8.772 (1.165) | 8.032 (1.146)
  Non-Smokers: number analyzed (Participants) | 27 | 28
  Non-Smokers | 10.575 (1.851) | 8.352 (1.676)
  Smokers: number analyzed (Participants) | 41 | 40
  Smokers | 6.969 (1.713) | 7.712 (1.563)

3. Primary Outcome: Self-report Weekly Smoking Craving
Description: Questionnaire of smoking urges (QSU). It has 32 questions that range from 1 to 7, there are 8 questions per sub-scale. The total range is 32 to 224. Each sub-scale ranges from 8- 56, with a higher score indicating higher craving.
Time Frame: 12 weeks
Population: Smokers only
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mecamylamine | Placebo
Number analyzed (Participants) | 41 | 40
units on a scale
  Desire to Smoke | 27.741 (1.311) | 28.047 (1.442)
  Anticipation of a positive outcome | 28.705 (1.718) | 28.273 (1.857)
  Relief | 22.557 (1.604) | 24.032 (1.730)
  Intention to smoke | 31.108 (1.793) | 32.549 (1.946)

4. Primary Outcome: Self-report Average Number of Cigarettes Per Day
Description: self-report from only the smoking population for cigarettes per day
Time Frame: 12 weeks
Population: only smokers
Measure: Mean (Standard Error); unit: cigarettes
Arm/Group | Mecamylamine | Placebo
Number analyzed (Participants) | 41 | 40
cigarettes | 8.055 (1.163) | 10.681 (1.258)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events were screened for on a weekly basis. Symptom data were clustered into the following categories: gastrointestinal (GI), central nervous system (CNS), neurological (NE), musculoskeletal (MS), skin, ophthalmological (OPTH), cardio/pulmonary (CAR), and genito-urinary (GU).
Groups:
- Mecamylamine Smoker; Mecamylamine Non-Smoker: mecamylamine: mecamylamine 10mg/day
- Placebo Smoker; Placebo Non-Smoker: Placebo: Placebo
Arm/Group | Mecamylamine Smoker | Mecamylamine Non-Smoker | Placebo Smoker | Placebo Non-Smoker
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/27 | 0/40 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/41 | 0/27 | 1/40 | 1/28
Other Adverse Events (participants affected / at risk) | 41/41 | 27/27 | 40/40 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mecamylamine Smoker (N=41) | Mecamylamine Non-Smoker (N=27) | Placebo Smoker (N=40) | Placebo Non-Smoker (N=28)
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Psychotic Delusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mecamylamine Smoker (N=41) | Mecamylamine Non-Smoker (N=27) | Placebo Smoker (N=40) | Placebo Non-Smoker (N=28)
gastrointestinal symptoms (Gastrointestinal disorders) | 29 | 17 | 22 | 18
central nervous system symptoms (Nervous system disorders) | 31 | 17 | 19 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes